CLINICAL TRIAL: NCT01447953
Title: Activity and Life-role Targeted Pain Rehabilitation in Primary Health Care: a Randomized Controlled Trial
Brief Title: Activity and Life-role Targeted Pain Rehabilitation in Primary Health Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organizational changes in health care made further recruitment to the treatment options unpossible.
Sponsor: Uppsala University (Other)
Collaborators: Center for Clinical Research Dalarna, Sweden (Other); Dalarna County Council, Sweden (Other); REHSAM, Sweden (Unknown)
Responsible Party: Principal Investigator, Catharina Gustavsson, RPT PhD, Principal Investigator Registered Physical Therapist PhD, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALAR-2009RS
Record Dates: First submitted 2011-09-09; First posted 2011-10-06 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Musculoskeletal Neck Pain; Musculoskeletal Shoulder Pain
Keywords: Activity; disability; life-role; multimodal rehabilitation; primary health care; persistent pain; randomized controlled trial; Musculoskeletal back pain
MeSH Terms: conditions — Shoulder Pain; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activity targeted pain rehabilitation (Experimental): A new activity and life-role targeting pain rehabilitation program (ALAR) has been developed to reduce psychosocial barriers to rehabilitation progress, promote re-integration into life-role activities and facilitate return-to-work.
  Interventions: Other: Activity targeted pain rehabilitation
- Treatment as usual (Active Comparator): Usual treatment consisting of multimodal rehabilitation provided by multi-professional teams in primary health care in the County of Dalarna, Sweden.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Activity targeted pain rehabilitation — An activity and life-role targeting rehabilitation programme (ALAR) provided by one of the care givers in the multi-professional rehabilitation teams at each of the eight participating primary health care centres, by ten weekly 1-hour treatment sessions.
  Arms: Activity targeted pain rehabilitation
Other: Treatment as usual — Usual treatment with type of treatment modalities, number, frequency and duration of visits according to the judgement of the muli-professional teams at each primary health care centre.
  Arms: Treatment as usual

SUMMARY:
The primary goal of the Swedish national rehabilitation plan on pain is to reduce disability and facilitate return-to-work. However, there is a lack of treatment strategies that effectively target and affect return-to-work and reduce sickness absence, and that in addition are sufficiently easy and feasible to administer in primary care. A new activity and life-role targeting rehabilitation program (ALAR) has been developed to reduce psychosocial barriers to rehabilitation progress, promote re-integration into life-role activities and facilitate return-to-work. The program will be implemented and provided as one of the pain treatment modalities available through multi-professional teams in primary care in one Swedish county. This study aims to evaluate the effect of an activity and life-role targeting pain rehabilitation program on the outcome variables return-to-work and sickness absence.

DETAILED DESCRIPTION:
The primary goal of the Swedish national rehabilitation plan on pain is to reduce disability and facilitate return-to-work. However, there is a lack of treatment strategies that effectively target and affect return-to-work and reduce sickness absence, and that in addition are sufficiently easy and feasible to administer in primary care. A new activity and life-role targeting rehabilitation program (ALAR) has been developed to reduce psychosocial barriers to rehabilitation progress, promote re-integration into life-role activities and facilitate return-to-work. The program will be implemented and provided as one of the pain treatment modalities available through multi-professional teams in primary care in one Swedish county. This study aims to evaluate the effect of an activity and life-role targeting pain rehabilitation program on the outcome variables return-to-work and sickness absence.

Patients seeking care due to disabling back, neck or shoulder pain at seven primary health care units in the County of Dalarna, Sweden, was randomly allocated to ALAR or usual multimodal rehabilitation. Between and within-group differences on return-to-work, sickness absence and disability will be evaluated at 10 weeks, six months, one and two years post-treatment.

The enrollment of patients was ended on preterm in june 2013. Due to changes in the organization in primary health care it was no longer possible to ensure that treatment arms could be delivered as intended. Data collection up to 1-year follow-up is completed. Data from longterm follow-up at 2 years will be completed in june 2015. Data analyses and reporting of results is presently undertaken. The number of enrolled participants is not enough to reach statistical power. Thus, results will need to be interpreted with caution.

Still the results of this pragmatic study will be of importance for the planning of a full scale study to accurately evaluate the effects of ALAR, to be conducted in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Persons seeking primary health care due to back, neck or shoulder pain
* Aged 18 to 60 years
* Being on sick leave or disability compensation
* Able to understand, read and write Swedish

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of days of sickness absence from work | 6 months
  Number of days of sickness absence from work during a 3-month period preceding the baseline measurement and preceding each follow-up, and specified in percent of full-time work.
Number of days of sickness absence from work | 1 year
  Number of days of sickness absence from work during a 3-month period preceding the baseline measurement and preceding each follow-up, and specified in percent of full-time work.
Number of days of sickness absence from work | 2 years
  Number of days of sickness absence from work during a 3-month period preceding the baseline measurement and preceding each follow-up, and specified in percent of full-time work.

SECONDARY OUTCOMES:
Return-to-work after sickness absence | Before treatment (at baseline), with follow-ups at 6 months, 1 , 2 and 5 years after treatment (after baseline assessment)
  Number of participants that return to work after sickness absence, i.e. that were on sick leave before the study and that has returned to work after the study.
Disability | Before treatment (at baseline), with follow-ups at 6 months, 1 , 2 and 5 years after treatment (after baseline assessment)
  Pain-related disability according to Pain Disability Index (PDI).

CONTACTS AND LOCATIONS:
Locations (1):
- The County Council of Dalarna; Primary Health Care units, Falun, Sweden